## **Consent Form**



**NHS Foundation Trust** 

Comparison of Nasopharyngeal and Lower Oesophageal Temperatures

Under General Anaesthesia with an Endotracheal Tube with Leak

Name of Investigators: Dr Haberman / Dr Snoek / Dr Hume-Smith

Patient Identification Number:

| $1.\square$ I confirm that I have read and understand the information of the above study. I have had the opportunity to consider these answered satisfactorily. | | |
|---|---|---|
| $2.\Box$ I understand that participation is voluntary and that without giving any reason, without our medical care or le | | at any time |
| 3. I understand that relevant sections of my child's metudy may be looked at by regulatory authorities or represermission for these individuals to have access to these re | sentatives from the NHS T | _ |
| $4.\square$ I agree to take part in the above study | | |
| Name of child | | |
| Name of parent / legal representative | Signature | Date |
| Name of person taking consent | Signature | Date |
| Name of investigator (if applicable) | Signature | Date |